CLINICAL TRIAL: NCT04947176
Title: A Double Blind, Randomized, Single Center, Controlled, Two Arm Trial of Dietary C15:0 Supplementation in Young Adults at Risk for Metabolic Syndrome
Brief Title: C15:0 Supplementation in Young Adults at Risk for Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jeffrey B. Schwimmer, MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey B. Schwimmer, MD, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 201339
Record Dates: First submitted 2021-06-09; First posted 2021-07-01 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): 200mg of pentadecanoic acid (C15:0) supplementation in capsules form
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): Matching placebo in capsules form
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — 200mg C15:0 once daily
  Arms: Active
Other: Placebo — Matching placebo once daily
  Arms: Placebo

SUMMARY:
This study will determine changes in plasma C15:0 levels in young adults with BMI ≥ 25 in response to 12 weeks of daily oral C15:0 supplementation.

DETAILED DESCRIPTION:
Metabolic syndrome is a disturbance in how the body processes both carbohydrates and fats. This condition has become common in children and young adults, especially in association with excess body fat. People with metabolic syndrome are at increased risk for type 2 diabetes, cardiovascular disease, and nonalcoholic fatty liver disease (NAFLD). Diet is believed to play an important role in both developing and treating metabolic syndrome. Studies have shown that low dietary intake of a type of fats known as odd chain fatty acids is associated with a higher risk for each of the metabolic syndrome associated conditions of diabetes, heart disease, and liver disease. Supplementation with one specific odd chain fatty acid known as C15:0 has shown to decrease the effects of metabolic syndrome in both cellular and animal models. In people, the epidemiology of consumption of C15:0 in the diet is consistent with this belief. However, clinical trials have yet to be done with supplemental C15:0. This study is a pilot study of C15:0 supplementation in a group of young adults at risk for metabolic syndrome. The study will determine how well supplementation with C15:0 daily for 12 weeks is able to raise levels of C15:0 in the blood when compared to placebo. The study will also look for signs that increasing blood levels of C15:0 leads to changes in physiology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 25 years
* Body Mass Index ≥ 25 Kg/m2

Exclusion Criteria:

* Reported habitual dietary intake of C15:0 that consistently exceeds 250 mg per day
* Significant alcohol consumption (average consumption >1 drink/day for females, >2 drink/day for males or episodes of binge drinking >5 drinks/day)
* Inability to swallow capsules
* Type 1 or Type 2 Diabetes
* Liver Cirrhosis
* Pregnancy
* Body weight greater than 125 kg at screening
* LDL-cholesterol > 160 mg/dL
* Triglycerides > 500 mg/dL
* Hemoglobin < 10.0 gm/dL
* Current Omega 3 Fatty Acid supplement usage
* Current use of Statin medications
* Any other condition which, in the opinion of the investigator, would impede compliance or hinder completion of the study
* Patients who are currently enrolled in a clinical trial or who received an investigational study drug within 180 days of screening.
* Subjects who are not able or willing to comply with the protocol or have any other condition that would impede compliance or hinder completion of the study, in the opinion of the investigator.
* Failure to give informed consent

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma C15:0 levels | Baseline to 12 weeks
  To determine changes in plasma C15:0 levels in response to daily supplementation of C15:

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline to 12 weeks
  To assess safety and tolerability of C15:0 supplementation as measured by number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Change in Weight | Baseline to 12 weeks
  Change in Weight (kg)
Change in BMI | Baseline to 12 weeks
  Change in BMI (kg/m^2)
Change in serum alanine aminotransferase | Baseline to 12 weeks
  Change in serum alanine aminotransferase (U/L)
Change in serum aspartate aminotransferase | Baseline to 12 weeks
  Change in serum aspartate aminotransferase (U/L)
Change in serum glutamyl transpeptidase | Baseline to 12 weeks
  Change in serum glutamyl transpeptidase (U/L)
Change in serum total cholesterol | Baseline to 12 weeks
  Change in serum total cholesterol (mg/dL)
Change in serum LDL-cholesterol | Baseline to 12 weeks
  Change in serum LDL-cholesterol (mg/dL)
Change in serum HDL-cholesterol | Baseline to 12 weeks
  Change in serum HDL-cholesterol (mg/dL)
Change in High Sensitivity C-reactive protein | Baseline to 12 weeks
  Change in High Sensitivity C-reactive protein (mg/L)
Change in serum glucose | Baseline to 12 weeks
  Change in serum glucose (mg/dL)
Change in serum insulin | Baseline to 12 weeks
  Change in serum insulin (μIU/mL)
Change in hemoglobin | Baseline to 12 weeks
  Change in hemoglobin (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Schwimmer, MD, Principal Investigator — UC San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Robinson MK, Lee E, Ugalde-Nicalo PA, Skonieczny JW, Chun LF, Newton KP, Schwimmer JB. Pentadecanoic Acid Supplementation in Young Adults with Overweight and Obesity: A Randomized Controlled Trial. J Nutr. 2024 Sep;154(9):2763-2771. doi: 10.1016/j.tjnut.2024.07.030. Epub 2024 Jul 26. PMID 39069269